CLINICAL TRIAL: NCT02951260
Title: The Effects of Metformin on Self-selected Exercise Intensity, Physical Fitness and Exercise-induced AMPK-activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Kristian Karstoft, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H- 16032037
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): 17 days metformin treatment
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): 17 days placebo treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — 17 days treatment with metformin
  Arms: Metformin
Other: Placebo — 17 days treatment with placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential interaction between metformin and exercise in order to optimize clinical guidelines for treatment of T2D.

DETAILED DESCRIPTION:
Physical activity is a first line treatment for patients with type 2 diabetes (T2D ), however, the vast majority of patients with T2D do not achieve satisfying glycemic control with physical activity alone, which is why pharmacological treatment with metformin is most often initiated. It is known that metformin and exercise both activates AMPK, which results in many different metabolic effects. Because of this similarity, an interaction between metformin and exercise is plausible, but knowledge in the area is sparse. With this study the investigators aim to look at the individual and combined effects of metformin and exercise in order to investigate whether an interaction occur. An Interaction will have tremendous clinical importance for patients with T2D given current guidelines where the vast majority of these patients are recommended both exercise and metformin treatment.

The investigators hypothesize that metformin treatment reduces self-selected exercise intensity, which may be explained via decreased mitochondrial complex 1 function, increased blood lactate levels, heart rate and RPE during exercise. Furthermore exercise-induced AMPK-activation is reduced with metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* male
* HbA1c < 39 mmol/l
* BMI < 25
* structured physical activity < = 150 min/week
* apparently healthy

Exclusion Criteria:

* smoking
* daily pharmaceutical treatment
* contraindication to increased levels of physical activity
* ALAT/ASAT elevated 3 times above upper normal values
* renal insufficiency (eGFR < 60 ml/min)
* prior history of lactic acidosis

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Overall aerobic work performed during an exercise bout with self-selected intensity | Total oxygen consumption (L O2) during a 45 min ergometer cycling bout with self-selected intensity

SECONDARY OUTCOMES:
External work performed during an exercise bout with self-selected intensity | Total work produced (kJ) during a 45 min ergometer cycling bout with self-selected intensity
Rate of perceived exertion during an exercise bout with fixed intensity | Mean rate of perceived exertion (Borg scale) during a 45 min ergometer cycling bout with fixed intensity
blood lactate during an exercise bout with fixed intensity | Mean blood lactate (mmol/l) during a 45 min ergometer cycling bout with fixed intensity
Heartrate during an exercise bout with fixed intensity | Mean heart rate (bpm) during a 45 min ergometer cycling bout with fixed intensity
Respiratory exchange ratio during an exercise bout with fixed intensity | Mean VCO2/VO2 during a 45 min ergometer cycling bout with fixed intensity
Physical fitness (VO2max) | maximal oxygen consumption (L/min) during a VO2 max test

OTHER OUTCOMES:
AMPK-activation in skeletal muscle during an exercise bout with fixed intensity | change in exercise induced AMPK-activation after compared to before a 45 min ergometer cycling bout with self-selected intensity
Oxidative phosphorylation in skeletal muscle fibers | Mitochondrial Complex I respiration in skeletal muscle tissue after 17 days of metformin/placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, PhD, Principal Investigator — Center for aktiv sundhed, Rigshospitalet
Locations (1):
- Center for aktiv sundhed, Copenhagen, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pilmark NS, Oberholzer L, Halling JF, Kristensen JM, Bonding CP, Elkjaer I, Lyngbaek M, Elster G, Siebenmann C, Holm NFR, Birk JB, Larsen EL, Lundby AM, Wojtaszewski J, Pilegaard H, Poulsen HE, Pedersen BK, Hansen KB, Karstoft K. Skeletal muscle adaptations to exercise are not influenced by metformin treatment in humans: secondary analyses of 2 randomized, clinical trials. Appl Physiol Nutr Metab. 2022 Mar;47(3):309-320. doi: 10.1139/apnm-2021-0194. Epub 2021 Nov 16. PMID 34784247